CLINICAL TRIAL: NCT02596542
Title: Cold Water Immersion as a Strategy to Promote Post-exercise Recovery in Healthy Young Men
Brief Title: Cold Water Immersion and Recovery
Acronym: CWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Lex Verdijk, Assistant Professor, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METC 153038
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Post-exercise Cold Water Immersion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Water temperature (Experimental)
  Interventions: Other: Water immersion

INTERVENTIONS:
Other: Water immersion — Different temperatures of cold water immersion will be assessed

SUMMARY:
Cold-water immersion (CWI) is a frequently applied strategy to accelerate post-exercise recovery in both recreational as well as professional athletes. However, the effect of repeated post-exercise CWI on other recovery strategies remains unclear.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Aged between 18-35 years
* Healthy, recreationally active
* BMI < 25 kg/m2
* The ability to comply with the protocol (i.e. the set-up for the CWI is designed for subjects that are at least 1.70 m or taller).

Exclusion Criteria:

* Smoking
* Allergies to milk proteins (whey or casein)
* Female
* Arthritic conditions
* A history of neuromuscular problems
* Recent (<1 y) participation in amino acid tracer studies
* Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Individuals with GI diseases

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis (expressed as fractional synthetic rate (FSR in %/h) | 2 weeks

SECONDARY OUTCOMES:
Muscle temperature (expressed as degrees celsius) | 1 day
Glycogen concentration (expressed as micromol glycosol units*g dry wt) | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SHM, Trommelen J, Kouw IWK, Holwerda AM, Pennings B, Groen BBL, Wall BT, Churchward-Venne TA, Horstman AMH, Koopman R, Burd NA, Fuchs CJ, Dirks ML, Res PT, Senden JMG, Steijns JMJM, de Groot LCPGM, Verdijk LB, van Loon LJC. Protein Type, Protein Dose, and Age Modulate Dietary Protein Digestion and Phenylalanine Absorption Kinetics and Plasma Phenylalanine Availability in Humans. J Nutr. 2020 Aug 1;150(8):2041-2050. doi: 10.1093/jn/nxaa024. PMID 32069356